CLINICAL TRIAL: NCT06909253
Title: Ravulizumab Treatment Outcomes in Patients With Generalized Myasthenia Gravis (gMG) Naive to Complement Inhibitors. Prospective, Multicenter, Non-interventional Study (MG-ARCADIA).
Brief Title: Ravulizumab Treatment Outcomes in Patients With Generalized Myasthenia Gravis
Acronym: MG-ARCADIA
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9281R00004
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Myasthenia Gravis, Generalized
Keywords: Ravulizumab; Generalized Myasthenia Gravis; gMG; observational
MeSH Terms: conditions — Myasthenia Gravis | interventions — ravulizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ravulizumab: Open-lable arm with gMG patients who received ravulizumab treatment in the frames of NDP in Poland.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Ravulizumab, concentrate for solution for infusion
  Other Names: Ultomiris

SUMMARY:
The Polish multicentre observational (non-interventional) study aiming to collect data on the management and clinical outcomes of patients with gMG that received ravulizumab.

DETAILED DESCRIPTION:
The Polish, prospective, multicenter, observational, cohort study designed to collect longitudinal data on the management and clinical outcomes of patients with gMG naive to complement inhibitors who received ravulizumab in the scope of routine clinical practice within the frames of National Drug Program (NDP) for up to 42 months (~ 6 months baseline and ~36 months follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged ≥18 years) patients with gMG, naive to complement inhibitors, receiving ravulizumab treatment in the frames of NDP in Poland.
* Patients willing to participate in the study and signed Informed Consent Form (ICF).
* Vaccination against N. meningitidis

Exclusion Criteria:

* Those who plan to participate in gMG clinical trial on/after the date of first ravulizumab infusion through NDP.
* Cognitive incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (aged ≥18 years) patients with gMG, naive to complement inhibitors, receiving ravulizumab treatment within the frames of NDP in Poland.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Myasthenia Gravis-Activities of Daily Living (MG-ADL) total score | at 6 month

SECONDARY OUTCOMES:
Change from baseline in Myasthenia Gravis-Activities of Daily Living (MG-ADL) total score | at month 12, 24, 36
Change from baseline in MG-ADL subcomponent scores | at month 6, 12, 24, 36
  Subcomponent scores - bulbar, limbs, respiratory, and ocular
Change from baseline in Myasthenia Gravis (MG) composite scale | at month 6, 12, 24, 36
Proportion of patients who achieved response | at month 6, 12, 24, 36
  Response - an improvement of ≥ 2 points in MG-ADL total score (proportion of patients with ≥ 3 improvement will be also presented)
Change in the Revised 15-Component Myasthenia Gravis Quality of Life (MG-QOL15r) score | at month 6, 12, 24, 36
Change from baseline in Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) | at month 6, 12, 24, 36
Change from baseline in Patient Global Impression of Change (PGI-C) | at month 6, 12, 24, 36
Change from baseline in Neuro-Qol Short Form v1.0 - Fatigue | at month 6, 12, 24, 36
Change from baseline in Patient Health Questionnaire - 9 (PHQ-9) | at month 6, 12, 24, 36

CONTACTS AND LOCATIONS:
Locations (10):
- Poland (10):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://vivli.org/